CLINICAL TRIAL: NCT05352971
Title: Multi-Site Validation of Ella Platform for Serum Nfl And GFAP Measures In Multiple Sclerosis Patients
Brief Title: Validation of Ella Platform for Serum Nfl And GFAP Measures In Multiple Sclerosis Patients
Acronym: Nf-Ella Loca
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: CIVI/2021/ET-02
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple sclerosis
  Interventions: Other: Biomarker quantification

INTERVENTIONS:
Other: Biomarker quantification — Patient blood samples will be tested on 2 different platforms

SUMMARY:
Serum neurofilament-light chain (NfL) and glial fibrillary acidic protein (GFAP) measured by single molecule array (SIMOA) are novel biomarkers of multiple sclerosis patients (MS) activity and progression. Its use is limited due to low availability and high costs. ELLA is a cheaper platform with increasing availability. Recently, we compared SIMOA and ELLA platforms to assess serum NfL levels in 203 MS patients from the OFSEP-HD study. There was a strong correlation (Spearman r = 0.86, p < 0.0001) between both platforms. As for SIMOA, serum NfL levels measured by ELLA were correlated with age and EDSS and were significantly higher in active MS, suggesting that these assays are equivalent and can be used in any center for routine care. However, the accuracy of local measures acquired with ELLA has not been determined. The aim os this study is to assess the concordance of multi-site ELLA instruments, accuracy of GFAP measures as compared to SIMOA, and the predictive value of NfL and GFAP measured by ELLA in MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the OFSEP HD cohort.
* At least one native (no thaw-freeze cycle) serum sample in local or in centralized Biological Resource Center

Exclusion Criteria:

* No bio-collection or insufficient sample volume
* No OFSEP minimal sheet at baseline

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MS from the OFSEP HD (NCT03603457) cohort.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Inter-laboratory reproducibility of neurofilament-light chain level measurements | Day 0
  Coefficients of variation will be calculated in 30 patients
Inter-laboratory repeatability of neurofilament-light chain level measurements | Day 0
  Serum from 3 patients with low, medium or high levels of NfL will be tested 10 times
Inter-laboratory reproducibility and repeatability of glial fibrillary acidic protein level measurements | Day 0
  Coefficients of variation will be calculated in 30 patients
Inter-laboratory repeatability of glial fibrillary acidic protein level measurements | Day 0
  Serum from 3 patients with low, medium or high levels of GFAP will be tested 10 times

SECONDARY OUTCOMES:
compare the GFAP values obtained using the ELLA and SIMOA platforms in MS patients | Day 0
  Intraclass concordance correlation coefficient and Passing-Bablock analysis calculated in 210 patients
to build a "global disease activity score" | Day 0
  Logistic regression to predict active multiple sclerosis
to build a "global disability score" | Day 0
  Logistic regression to predict Expanded Disability Status Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU de Nimes
Locations (10):
- France (10):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU Gui de Chauliac, Montpellier
  - CHU de Nantes,, Nantes
  - Centre Hospitalier Universitaire Pasteur 2, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU de Strasbourg, Strasbourg